CLINICAL TRIAL: NCT01346904
Title: The Central Nerve System Injury in Patients With Primary Open Angle Glaucoma
Brief Title: a 3.0T Magnetic Resonance Imaging Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: HONG ZHANG, Department of Opthalmology ,Tongji Hospital
Other Study IDs: POAG3243
Record Dates: First submitted 2011-05-02; First posted 2011-05-03 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Glaucomatous damage not only occurred to retinal ganglion cells in the eyes, but went across optic nerves, visual chiasm, lateral geniculate nucleus (LGN) and finally the visual cortex; the neural degenerations could be identified through the whole visual tract, which suggests the central nerve system may play a vital role in the progression of glaucoma. The investigators used MRI to investigate changes of visual pathway in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma diagnosed on the basis of glaucomatous optic disc cupping ratio (in particular, thinning of the inferior and/or superior rim, cup-to-disc ratio asymmetry of >0.2)
* matching glaucomatous visual field defects (European Glaucoma Society (2008) Perimetry )

Exclusion Criteria:

* optic neuropathy
* neurological disorder
* other diseases and use of systemic medications which affect optic nerve or the visual ﬁeld underwent complete eye examination and visual-field testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects recruited from the Department of Ophthalmology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology. Clinical ophthalmic assessments including measurement of visual acuities, intraocular pressure, slit-lamp microscopes and funduscopes examinations, cup-to-dick ratio (CDR) evaluation, visual field test [Octopus 101 Automated Perimeter, Haag-streit, Switzerland. Program G2], optical coherence tomography for retinal nerve fiber layer thickness(RNFLT) around the optic disk[Stratus OCT，Carl Zeiss Meditec, Dublin, CA .Scan Type :Fast RNFLT 3.4, Scan Length: 10.87mm].
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: HONG ZHANG, PHD, Study Chair — Tongji Hospital